CLINICAL TRIAL: NCT00131937
Title: A Phase II Study of Sorafenib (BAY 43-9006) in Recurrent Aggressive Non-Hodgkin's Lymphoma
Brief Title: Sorafenib Tosylate in Treating Patients With Recurrent Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00658; E1404 (Other: Eastern Cooperative Oncology Group); U10CA021115 (NIH)
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Results first posted 2015-09-03 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-07

CONDITIONS: Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Hepatosplenic T-cell Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib 400 mg PO twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with recurrent diffuse large B-cell non-Hodgkin's lymphoma. Sorafenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response rate of treatment with sorafenib (BAY43-9006) in patients with recurrent aggressive non-Hodgkin's lymphomas.

SECONDARY OBJECTIVES:

I. To evaluate the duration of response and progression free survival of treatment with BAY43-9006 in patients with recurrent aggressive Non-Hodgkin's Lymphomas.

II. To characterize the toxicity of treatment with BAY43-9006 in patients with recurrent aggressive Non-Hodgkin's Lymphomas.

III. To further characterize the pharmacokinetics properties of BAY43-9006 and assess influence of monooxygenases polymorphisms and multi-drug resistance transporter (MDR) on pharmacokinetics.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PLANNED ACCRUAL: 41 ACTUAL ACCRUAL: 14

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed recurrent de novo or transformed diffuse large B cell lymphoma (DLBCL) or one of its variants according to WHO classification (centroblastic, immunoblastic, T-cell/histiocyte rich and anaplastic variants)
* Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1
* Patients must have measurable disease as defined in section 6 assessed within 4 weeks of registration
* Patients must have failed one or more prior Non-Hodgkin lymphoma (NHL) chemotherapy or antibody therapy with curative intent; autologous stem cell transplant is permitted
* Leukocytes >= 2,000/mm^3
* Absolute neutrophil count >= 1,000/mm^3
* Platelets >= 75,000/ mm^3
* Total bilirubin =< 2.0 X normal institutional limits
* Aspartate Aminotransferase (AST) =< 2.5 X institutional upper limit of normal
* Alanine Aminotransferase (ALT) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits; creatinine clearance calculated or measured at >= 60 ml/min/1.73m^2 if creatinine level is above institutional limits
* The prothrombin time (PT)/international normalized ratio (INR) within Institutional limits of normal
* Patients with underlying hypertension as defined by blood pressures averaging greater than 140/90 on two separate clinic visits are eligible if hypertension has been controlled by standard nonpharmacologic and pharmacologic therapy
* Patients must be physically able to orally ingest tablets

Exclusion Criteria:

* Central nervous system (CNS) involvement
* Previously treated with Sorafenib (BAY 43-9006) or other small molecule targeted inhibitors of mitogen-activated protein kinase (MAPK) signaling intermediates or angiogenesis (e.g. bevacizumab)
* Progressed within 60 days of last therapy
* Prior allogeneic stem cell transplant
* Candidates for potentially curative therapy, such as hematopoietic stem cell transplantation (HSCT)
* Currently receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements
* Active HIV infection, because of possible pharmacokinetic interactions of anti-retroviral therapy with BAY43-9006
* Evidence of bleeding diathesis
* Currently taking the cytochrome P450 enzyme-inducing anti-epileptic drugs (phenytoin, carbamazepine and phenobarbital), rifampin or St. John's Wort
* Pregnant or Breast-feeding; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy. Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-10; Primary Completion 2011-09 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Horning, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Sorafenib): Patients receive oral sorafenib 400 mg PO twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  sorafenib tosylate: Given orally
Period: Overall Study
Arm/Group | Treatment (Sorafenib)
Started | 14
Completed | 0
Not Completed | 14
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Disease Progression | 7
Not completed — Alternative therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Sorafenib)
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 69.5 [38 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR) Rate
Description: Response was assessed using the criteria from International Workshop to Standardize Criteria for NHL (Cheson, 1999). OR=complete response(CR)+complete response/uncertain(CRu)+partial response(PR) CR: 1)Disappearance of clinical/radiographic evidence of disease (dz) and all dz-related B-symptoms; normalization of biochemical abnormalities attributed to NHL; 2)Lymph nodes and nodal masses regress to normal size; 3)Spleen, if enlarged before therapy, has decreased in size and is not palpable; 4)Complete resolution of lymphoma in bone marrow biopsy CRu: Meet criteria 1 and 3 above but with ≥1 of the followings. Residual dominant nodal mass >1.5 cm in greatest diameter that has decreased by >75%. Indeterminate bone marrow.
  PR: ≥50% decrease in SPD (sum of products of diameters) of 6 largest dominant nodes or nodal masses. No increase in size of liver or spleen. No unequivocal progression in nonmeasurable or nondominant sites. Splenic/hepatic nodules regress ≥50% in SPD. No new dz sites.
Time Frame: Assessed at the end of Cycle 2 and Cycle 6 (1 cycle = 28 days). Then every 3 months beginning Cycle 9 if patient is < 2 years from study entry, every 6 months if patient is 2-3 years from study entry, up to 3 years.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Groups:
- Treatment (Sorafenib): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  sorafenib tosylate: Given orally
Arm/Group | Treatment (Sorafenib)
Number analyzed (Participants) | 14
Proportion of participants | 0.07 [0.004 to 0.30]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first of progression, relapse or death from any cause. Per criteria from International Workshop to Standardize Criteria for NHL (Cheson, 1999), progression (for patients who have not responded) and relapse (for patients who responded) are defined as:
  1. Appearances of any new lesions/sites during or after therapy
  2. Increase of ≥50% in the SPD from nadir measurement of all involved dominant lymph nodes and liver/spleen nodules or unequivocal progression in any nonmeasurable disease or nondominant site
  3. Increase by ≥50% in greatest diameter from nadir measurement of any previously involved dominant node >1.0 cm in its short axis
Time Frame: Assessed after month 2 and month 6, then every 3 months if patient is < 2 years from study entry, every 6 months if patient is 2-3 years from study entry, up to 3 years
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Sorafenib)
Number analyzed (Participants) | 14
months | 2 [1 to 5]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study entry until death from any cause.
Time Frame: as for outcome 2
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Sorafenib)
Number analyzed (Participants) | 14
months | 9 [5 to 16]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Treatment (Sorafenib): All patients who received Sorafenib treatment.
Arm/Group | Treatment (Sorafenib)
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sorafenib) (N=14)
White blood cell decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Hypertension (Vascular disorders) | 1
Fatigue (General disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sorafenib) (N=14)
Allergic reaction (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 5
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Hypertension (Vascular disorders) | 7
Fatigue (General disorders) | 10
Weight loss (Investigations) | 1
Flushing (Vascular disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 8
Flatulence (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, spec (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 3
Musculoskeletal and connective tissue di (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The study did not meet pre-specified criteria for continuing to second stage accrual (at least one response among the first 12 eligible patients), and was therefore closed per protocol without full accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less